CLINICAL TRIAL: NCT04095143
Title: Ultrasound Markers of Organ Congestion in Severe Acute Kidney Injury
Acronym: ECHO-AKI
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Unity Health Toronto (Other); Sunnybrook Health Sciences Centre (Other); University of Kentucky (Other); University of Alberta (Other); Montreal Heart Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MP-02-2020-8578 (MP)
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Acute Kidney Injury; Fluid Overload; Ultrasonography
Keywords: Point-Of-Care ultrasound; Doppler; Major adverse kidney events; Portal flow pulsatility; IVC ultrasound; Cardiac ultrasound; Right ventricular failure; Intensive care
MeSH Terms: conditions — Acute Kidney Injury; Edema; Heart Failure | interventions — Ventricular Function, Left; Ventricular Function, Right

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- New onset of stage ≥2 acute kidney injury: Either:
  1. A ≥ 2-fold increase in serum creatinine OR
  2. A serum creatinine ≥ 354 μmol/L with evidence of a minimum increase of 27 μmol/L OR
  3. Urine output < 6.0 mL/kg over the preceding 12 hours OR
  4. Initiation of RRT for severe acute kidney injury less than 72 hours before recruitment
  Interventions: Diagnostic Test: Portal vein flow; Diagnostic Test: Intra-renal flow; Diagnostic Test: Hepatic vein flow; Diagnostic Test: Pulmonary B-lines; Diagnostic Test: Dimensions of the inferior vena cava; Diagnostic Test: Left ventricular function; Diagnostic Test: Right ventricular function

INTERVENTIONS:
Diagnostic Test: Portal vein flow — Doppler assessment performed on day 0, 3 and 7.
Diagnostic Test: Intra-renal flow — Doppler assessment performed on day 0, 3 and 7.
Diagnostic Test: Hepatic vein flow — Doppler assessment performed on day 0, 3 and 7.
Diagnostic Test: Pulmonary B-lines — Ultrasound assessment of performed on day 0, 3 and 7.
Diagnostic Test: Dimensions of the inferior vena cava — Ultrasound assessment of performed on day 0, 3 and 7.
Diagnostic Test: Left ventricular function — Ultrasound assessment of performed on day 0, 3 and 7.
Diagnostic Test: Right ventricular function — Ultrasound assessment of performed on day 0, 3 and 7.

SUMMARY:
Fluid overload is associated with adverse outcomes in patients with severe acute kidney injury. It remains unclear if fluid overload is merely a marker of disease severity or if organ congestion is a mediator of complications. Point-of-care ultrasound could be a modality used to assess organ congestion and its clinical implications. The objective of this study is to determine whether ultrasound markers of organ congestion are associated with major adverse kidney events in critically ill patients with severe acute kidney injury.

DETAILED DESCRIPTION:
Background: Fluid overload is associated with adverse outcomes in patients with severe acute kidney injury. It remains unclear if fluid overload is merely a marker of disease severity or if organ congestion is a direct mediator of complications. Point-of-care ultrasound could be a modality used to assess organ congestion and its clinical implications.

Objective: To determine whether ultrasound markers of organ congestions are associated with major adverse kidney events and other adverse clinical outcomes.

Study design: A cohort of critically ill patients with a new onset of severe acute kidney injury will undergo repeated ultrasound assessments to detect the presence of the following markers:

* Portal flow pulsatility on pulse-wave Doppler
* Discontinuous intra-renal venous flow on pulse-wave Doppler
* Abnormal hepatic vein waveform on pulse wave Doppler
* Presence of pulmonary B-line artifacts on 2D lung ultrasound
* Presence of dilated and non-collapsible inferior vena cava on 2D ultrasound
* Presence of systolic right ventricular dysfunction
* Presence of systolic left ventricular dysfunction

Clinical outcomes will be collected for up to 90 days after recruitment.

Perspective: An approach targeting the resolution of organ congestion might improve the prognosis in patients with severe acute kidney injury. Identifying clinically relevant markers of organ congestion is a precursor to the design of future interventional trials investigating personalized fluid balance management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admitted to the ICU
* Women with serum creatinine ≥ 100 µmol/L and men with serum creatinine ≥ 130 µmol/L
* Severe acute kidney injury (AKI) defined either: A ≥ 2-fold increase in serum creatinine from a known pre-morbid baseline or during the current hospitalization OR achievement of a serum creatinine ≥ 354 µmol/L with evidence of a minimum increase of 27 µmol/L from pre-morbid baseline or during the current hospitalization OR Urine output < 6.0 mL/kg over the preceding 12 hours OR initiation of renal replacement therapy (RRT) for severe AKI initiated less than 72 hours before recruitment.

Exclusion Criteria:

* Lack of commitment to provide RRT as part of limitation of ongoing life support. (Operational definition: Critical care team has deemed the patient not to be eligible for escalation of life support, including the initiation of RRT, or substitute decision makers have declined offer of same.)
* Known pre-hospitalization advanced chronic kidney disease, defined by an estimated glomerular filtration rate < 20 mL/min/1.73 m2 in a patient who is not on chronic RRT. (Operational definition: The coordinator will review all documented serum creatinine values within 365 days prior to the date of admission for the current hospitalization. The value closest to the admission date will be considered as the "baseline" and will be used to calculate the corresponding estimated glomerular filtration rate using an online calculator. A value of < 20 mL/min/1.73 m2 derived from the CKD-EPI equation will be grounds for exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult patients with severe acute kidney injury
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with major adverse kidney events at 30 days | 30 days
  Either death, receipt of renal replacement therapy or sustained loss of kidney function (new onset of estimated glomerular filtration rate (eGFR) < 60 or, if pre-existing eGFR < 60, 25% or greater decline in eGFR)

SECONDARY OUTCOMES:
Rate of in-hospital death | 30 days
  All cause mortality during hospital stay
Number of participants with renal replacement therapy dependence at 30 days | 30 days
  Receipt of renal replacement therapy at 30 days from enrollment
Number of participants with sustained loss of kidney function at 30 days | 30 days
  New onset of estimated glomerular filtration rate (eGFR) < 60 or, if pre-existing eGFR < 60, 25% or greater decline in eGFR)
Ventilation-free days through day 30 | 30 days
  A ventilator-free day will be defined as the receipt of < 2 hours of either invasive or non-invasive ventilation within a 24-hour period.
Intensive care unit (ICU)-free days through day 30 | 30 days
  An ICU-free day will be defined as admission to an ICU for < 2 hours within a 24 hours period.
Vasopressor-free days though day 30 | 30 days
  Vasopressor will include norepinephrine, epinephrine, vasopressin and phenylephrin
Number of participants with major adverse kidney events at 90 days | 90 days
  Either death, receipt of renal replacement therapy or sustained loss of kidney function (estimated glomerular filtration rate (eGFR) < 60 or, if pre-existing eGFR < 60, 25% or greater decline in eGFR)
Rate of death at 90 days | 90 days
  All cause mortality at 90 days
Estimated glomerular filtration rate at 90 days | 90 days
  Calculated with the CKD-EPI equation (92) with serum creatinine from a sample drawn as close as possible to Day 90.

OTHER OUTCOMES:
Hemodynamic instability during renal replacement therapy | 7 days
  Intradialytic hypotension (MAP<65 mmHg) requiring one or more of the following interventions: interruption of fluid removal, introduction of norepinephrine or increase in its dose of more than 25%, administration of volume expansion or interruption of RRT within 8 hours after initiating net negative fluid balance.

CONTACTS AND LOCATIONS:
Overall Officials: William Beaubien-Souligny, MD, Principal Investigator — CHUM
Locations (6):
- University of Kentucky, Lexington, Kentucky, United States
- Canada (5):
  - University of Alberta, Edmonton, Alberta
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - St. Michael's hospital, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided